CLINICAL TRIAL: NCT05666700
Title: CAR-T Cell Therapy in RelApsed/Refractory Myeloma With ExtrameduLlary Disease - an in Vivo Imaging and Molecular Monitoring Study
Acronym: CARAMEL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/015
Record Dates: First submitted 2022-12-04; First posted 2022-12-28 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Extramedullary Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cilta-cel (Experimental)
  Interventions: Biological: Combination Product: JNJ-68284528 (Cilta-cel) & 64Cu SPION dual PET-MR imaging agent

INTERVENTIONS:
Biological: Combination Product: JNJ-68284528 (Cilta-cel) & 64Cu SPION dual PET-MR imaging agent — Cilta-cel is a cellular immunotherapy derived from autologous CD3+ T-cells that have undergone ex vivo modification to target B-Cell Maturation Antigen (BCMA) on the surface of plasma cells. Cilta-cel will be administered as two IV infusions, ≥70% unlabeled and ≤30% labelled. The dose will be based on the patient's weight (kg) at apheresis

SUMMARY:
This clinical trial will investigate the in vivo trafficking of cilta-cel in extramedullary myeloma using 64Cu Super Paramagnetic Iron Oxide Nanoparticle (64Cu SPION) and Positron Emission Tomography-Magnetic Resonance Imaging (PET-MRI)

DETAILED DESCRIPTION:
This a Phase Ib exploratory study designed to investigate the in vivo trafficking of cilta-cel in extramedullary myeloma (EMM) using 64Cu SPION nanoparticles and PET-MRI imaging. It is planned that 10-30% of clinical dose of target number of cilta-cel will be labelled. The target number cilta-cel has been chosen based on the previous first in humans (FIH) study. The rationale to label of cilta-cel in the range of ≤30% is to ensure that reasonable positron emission tomography (PET) and magnetic resonance (MR) imaging quality by increasing the relative labelling dose, in the case low cell numbers are obtained. Additionally, the selected range is chosen to limit cellular toxicity and radiation exposure to the patient from the labelled cells. The unlabeled and labelled dose will be administered as scheduled by a two-part intravenous infusion in which the labelled cells are administered no later than 4hrs after the unlabeled infusion

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria for study entry:

1. Patient has provided written informed consent
2. Patient is >18 years of age at the time of consent
3. Patient has a documented diagnosis of MM according to the IMWG diagnostic criteria (Appendix 1)
4. Measurable extramedullary disease by any imaging modality (at least one site of disease ≥1cm that has never received radiotherapy or has progressed following radiotherapy). Presence of biochemical measurable disease is not required
5. Have received at least 2 prior lines of therapy including a PTI and an IMiD. Patient must have undergone at least 1 complete cycle of treatment for each line of therapy, unless PD was the best response to the line of therapy (Appendix 2) Note: induction with or without haematopoietic stem cell transplant, consolidation and maintenance therapy is considered a single line of therapy.
6. Have an ECOG Performance Status score of 0 or 1 (Appendix 3)
7. Have a life expectancy of ≥3 months, as judged by the Investigator
8. Able to undergo apheresis for mononuclear cell collection
9. Have clinical laboratory values meeting the following criteria within 7 days prior to registration (enrolment):

   * Haemoglobin ≥80g/L (recombinant human erythropoietin use is permitted)
   * ANC ≥1 × 109/L (prior growth factor support is permitted but must be without support in the 7 days prior to the laboratory test)
   * Platelet count ≥50 × 109/L
   * Absolute lymphocyte count ≥0.3 × 109/L
   * AST ≤3.0× ULN
   * ALT ≤3.0× ULN
   * Total bilirubin ≤2.0× ULN; except in patients with congenital bilirubinaemia, such as Gilbert's syndrome (in which case direct bilirubin ≤2.0× ULN is required)
   * Calculated CrCl ≥40mL/min calculated by the Cockcroft-Gault formula (Appendix 4), nuclear medicine assessment or a 24-hour urine collection
10. When a woman is of childbearing potential, the patient must commit either to abstaining continuously from heterosexual intercourse or agree to practice 2 methods of reliable birth control simultaneously. Where one of the methods is highly effective method of contraception (failure rate of <1% per year when used consistently and correctly; see examples below) and one other effective method (i.e., male latex or synthetic condom, diaphragm, or cervical cap) and patient must agree to remain on both methods from the time of signing the PICF until at least 1 year after receiving a cilta-cel infusion (Appendix 5). Reliable contraception is indicated even where there has been a history of infertility, unless it is due to hysterectomy. WOCBP should be referred to a qualified provider of contraceptive methods, if needed. Examples of highly effective contraceptives include:

    * User-independent methods: 1) implantable progestogen-only hormone contraception associated with inhibition of ovulation; 2) intrauterine device; intrauterine hormone-releasing system; 3) vasectomised partner
    * User-dependent method: progestogen-only hormone contraception associated with inhibition of ovulation (oral or injectable)
11. A man must commit either to abstaining continuously from heterosexual intercourse or a man who is sexually active with a WOCBP or a pregnant woman must agree to use a barrier method of contraception (e.g., latex or synthetic condom with spermicidal foam/gel/film/cream/suppository) from the time of signing the PICF until at least 1 year after receiving a cilta-cel, even if they have undergone a successful vasectomy
12. Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, until at least 1 year after receiving a cilta-cel infusion
13. Patient must be willing and able to adhere to the following lifestyle restrictions during the study to be eligible for participation:

    * Refer to Section 8.6.3, Prohibited Therapies for details regarding prohibited and restricted therapy during the study
    * Agree to follow all requirements that must be met during the study as noted in the Inclusion and Exclusion Criteria (e.g., contraceptive requirements)

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Known nickel or Pd sensitivity
2. Weight >105 Kg and/or height >185 cm
3. Known claustrophobia
4. Prior treatment with CAR-T therapy directed at any target
5. Received a cumulative dose of corticosteroids equivalent to ≥70mg of prednisone within the 7 days prior to planned apheresis
6. Any prior therapy that is targeted to BCMA
7. Vaccination with an investigational vaccine or live attenuated vaccine (except for COVID-19) within 4 weeks prior to planned conditioning
8. Patient received any anti-tumour therapy as follows, prior to planned apheresis:

   * Targeted therapy, epigenetic therapy, or treatment with an investigational drug or use of an invasive investigational medical device within 14 days or at least 5 half-lives, whichever is less
   * Investigational vaccine within 4 weeks
   * Monoclonal antibody treatment within 21 days
   * Cytotoxic therapy within 14 days
   * Radiotherapy within 14 days. However, if the radiation is given for palliative purposes and the radiation portal covered ≤5% of the bone marrow reserve, the patient is eligible irrespective of the end date of radiotherapy
9. Active malignancies (i.e., progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. The only allowed exceptions are:

   * Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured
   * Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured
   * Non-invasive cervical cancer treated within the last 24 months that is considered completely cured
   * Localised prostate cancer (N0M0):

     * With a Gleason score of ≤6, treated within the last 24 months or untreated and under surveillance
     * With a Gleason score of 3+4 that has been treated more than 6 months prior to full study screening and considered to have a very low risk of recurrence, or
     * History of localised prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence
   * Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localised breast cancer and receiving anti-hormonal agents and considered to have a very low risk of recurrence
   * Malignancy that is considered cured with minimal risk of recurrence
10. Plasma cell leukaemia at the time of screening (>2.0 x 109/L plasma cells by standard differential), Waldenström's macroglobulinaemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloid light-chain amyloidosis
11. Contraindications or known life-threatening allergies, hypersensitivity, or intolerance to any of the study treatments (if known) or any of their excipients, including boron, mannitol, and dimethyl sulfoxide (refer to IB), or local product prescribing information for complete lists of excipients
12. Pregnant or breast-feeding or planning to become pregnant while enrolled in this study or within 1 year after receiving cilta-cel infusion
13. Plans to father a child while enrolled in this study or within 1 year after receiving cilta-cel infusion
14. Stroke or seizure within 6 months prior to signing PICF
15. Received either of the following:

    * An allogenic stem cell transplant within 6 months before planned apheresis. Patients who received an allogeneic transplant must have stopped all immunosuppressive medications for 6 weeks without signs of graft-versus-host disease. Patients with active graft-versus-host disease are excluded
    * An ASCT ≤12 weeks before planned apheresis
16. Known active, or prior history of, CNS involvement or exhibits clinical signs of meningeal involvement of MM
17. Any of the following criterion related to infectious diseases:

    * Seropositive for HIV
    * Hepatitis B infection: In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status (Appendix 6)
    * Hepatitis C infection (defined as anti -HCV antibody positive or HCV-RNA positive) or known to have a history of hepatitis C NOTE: For patients with positive HCV antibody due to prior resolved disease can be enrolled, only if a confirmatory HCV RNA test is undetectable. For patients with known history of HCV infection, confirmation of sustained virologic response is required for study eligibility, defined as undetectable HCV RNA ≥24 weeks after completion of antiviral therapy.
18. Serious underlying medical or psychiatric condition or disease, that is likely to interfere with study procedures or results, or that in the opinion of the Investigator would constitute a hazard for participating in this study, such as:

    * Requirement of continuous supplemental oxygen
    * Evidence of active viral or bacterial infection, requiring systemic antimicrobial therapy, or uncontrolled systemic fungal infection
    * Active autoimmune disease
    * Overt clinical evidence of dementia or altered mental status
    * Any history of Parkinson's disease or other neurodegenerative disorder
    * Clinically significant cardiac conditions, such as:

      * NYHA Class III or IV congestive heart failure (Appendix 7) Short title: CARAMEL Page 60 of 128 Version: 1.0 Date: 17th November 2022
      * Myocardial infarction or coronary-artery-bypass graft ≤6 months prior to planned apheresis
      * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
      * History of severe non-ischemic cardiomyopathy
      * Impaired cardiac function (LVEF <45%) as assessed by ECHO or MUGA scan performed ≤8 weeks before planned apheresis
19. Major operations or surgical procedures within 2 weeks prior to bridging therapy, or has surgery planned during the study or within 2 weeks after study treatment administration Note: patients with planned surgical procedures to be conducted under local anaesthesia may participate.
20. Frailty index of ≥ 2 according to Myeloma Geriatric Assessment score (Appendix 8)
21. Any issue that would impair the ability of the patient to receive or tolerate the planned treatment, to understand informed consent or any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To determine the utility of 64Cu SPION labelling for in vivo real time monitoring of trafficking of anti-BCMA Chimeric Antigen Receptor T-Cell (CAR-T) cells in Relapsed/ Refractory (RR) EMM. | assessed up to one month (first month after infusion)
  Detectable cells by PET assessed by the Deauville score >3

SECONDARY OUTCOMES:
Safety of 64Cu SPION labelled cilta-cel for EMM | From date of signing consent until study completion, assessed up to approximately 31 months
  Incidence, nature and severity of adverse events (AEs) according to Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) and 2019 American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria for cytokine release syndrome (CRS) and neurotoxicity, Serious Adverse Events (SAE), and Adverse Events of special interest (AESI)
Complete response rate (CRR) by International Myeloma Working Group (IMWG) criteria | assessed up to approximately 13 months
  Using IMWG criteria
Overall response rate (ORR) by IMWG criteria | assessed up to approximately 13 months
  Using IMWG criteria
Minimal residual disease response by Adaptive ClonoSeq assay | assessed up to approximately 13 months
  on ctDNA at Day +1, Day +28, 12 weeks, 24 weeks, and 52 weeks post Day +28 and on Bone Marrow Aspirate (BMA) at Day +28 and at suspected CR
Duration of Response by IMWG criteria | assessed up to approximately 13 months
  Defined as time from first response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR) to time to progressive disease (PD)
Progression free survival, defined as time from study enrolment until biochemical, radiological and/or clinical PD or death, according to IMWG criteria | assessed up to approximately 13 months
  by IMWG criteria
Overall survival (OR) | assessed up to approximately 31 months
  defined as time from study enrolment to death

CONTACTS AND LOCATIONS:
Overall Officials: Simon Harrison, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No